CLINICAL TRIAL: NCT02249494
Title: Nutritional Recommendations for Hypertension: Development of Mobile Application for Improve Knowledge in Lifestyle Modification for Primary Care Physicians
Brief Title: Mobile Application to Improve Nutritional Counseling Provided by Primary Care Physicians for Hypertension.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-0258
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension
Keywords: Nutritional Knowledge; Nutritional Counseling
MeSH Terms: conditions — Hypertension | interventions — Telemedicine; Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smartphone (mobile app) & telehealth (Experimental): Participants will install and use a mobile application designed to provide nutritional recommendations for hypertensive patients. These recommendations will be based on the DASH diet guidelines appropriate to patient profile: consumption of whole grains, fruits, vegetables, milk or low fat dairy products, lean meats, poultry and fish, nuts, seeds and legumes, amount of fats, oils and sweets, as well as guidelines for salt intake and alcohol. The call service will be offered by the Center for Telehealth Rio Grande do Sul to answer clinic questions with qualified staff and in real time. All physicians who work in Primary Health Care in Brazil can use this call center when they have questions about diagnosis and management of their patients.
  Interventions: Other: telehealth; Other: nutritional counseling; Device: smartphone (mobile app)
- nutritional counseling & telehealth (Placebo Comparator): Physicians who are enrolled for this group will continue performing routine nutritional counseling in their clinical practice. The call service will be offered by the Center for Telehealth Rio Grande do Sul to answer clinic questions with qualified staff and in real time. All physicians who work in Primary Health Care in Brazil can use this call service when they have questions about diagnosis and management of their patients.
  Interventions: Other: telehealth; Other: nutritional counseling

INTERVENTIONS:
Other: telehealth — Use the call service offered by the Center for Telehealth Rio Grande do Sul to answer clinic questions with qualified staff and in real time. All physicians who work in Primary Health Care in Brazil can call when they have questions about diagnosis and management of their patients.
Other: nutritional counseling — Performing routine nutritional counseling in their clinical practice
Device: smartphone (mobile app) — Mobile app, designed to provide nutritional recommendations for hypertensive patients, will be use. The recommendations will be based on the DASH diet guidelines appropriate to the patient profile: consumption of whole grains, fruits, vegetables, milk or low fat dairy products, lean meats, poultry and fish, nuts, seeds and legumes, amount of fats, oils and sweets, as well as guidelines for salt intake and alcohol.
  Arms: Smartphone (mobile app) & telehealth

SUMMARY:
The purpose of this study is to investigate whether the use of a mobile app could improve knowledge and practice in nutrition counseling performed by primary care physicians in Brazil.

DETAILED DESCRIPTION:
To optimize the nutritional care in the context of the limitations of available time and knowledge in medical practice, the present study proposes to develop a tool of nutritional guidelines for hypertension, easily accessible, based on evidence, and then evaluate its use among primary care physicians registered in a center telehealth. The use of the mobile application tool will aim to improve the nutritional counseling, helping with prevention of other chronic diseases in primary care context.

ELIGIBILITY:
Inclusion Criteria:

* primary care physicians registered in TelessaúdeRS (Center for Telehealth)
* primary care physicians who use smartphone or tablet

Exclusion Criteria:

* not to work in primary care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in score of knowledge and ability related to nutritional care. | 30 days
  For each correct answer, participant will get one point on the knowledge test and for each incorrect answer will get 0. Thus, possible scores will range from 69 to 0. Data based on questions about the abilities will be summarized in a qualitative ranking.

CONTACTS AND LOCATIONS:
Overall Officials: Erno Harzheim, doctor, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Núcleo de Telessaúde Técnico-Científico do Rio Grande do Sul. Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Gadenz SD, Harzheim E, Rados DRV, Castro SMJ, Drehmer M. Mobile Application Increased Nutrition Knowledge Among Brazilian Physicians. J Nutr Educ Behav. 2024 Feb;56(2):92-99. doi: 10.1016/j.jneb.2023.11.001. Epub 2023 Dec 21. PMID 38127014